CLINICAL TRIAL: NCT01624012
Title: Non-invasive Ventilation With Neurally Adjusted Ventilatory Assist (NIV NAVA) Versus Nasal Continuous Airway Pressure (NCPAP) in Premature Infants
Brief Title: Non-invasive Ventilation With Neurally Adjusted Ventilatory Assist Versus Nasal Continuous Airway Pressure in Premature Infants
Acronym: NIV NAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Merja Ålander, Principal investigator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EETTMK:23/2011
Record Dates: First submitted 2012-06-04; First posted 2012-06-20 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Respiratory Distress Syndrome (RDS) of Neonate
Keywords: NIV NAVA; non-invasive ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIV NAVA (Active Comparator): Noninvasive ventilation in this group is practiced with NIV NAVA
  Interventions: Device: NIV NAVA
- ncpap (Active Comparator): Patients randomized to this arm will receive noninvasive ventilation with continuous nasal CPAP as routinely in neonatal intensive care unit.
  Interventions: Device: Nasal continuous positive airway pressure

INTERVENTIONS:
Device: NIV NAVA — Non invasive ventilation with neurally adjusted ventilatory assist
  Arms: NIV NAVA
Device: Nasal continuous positive airway pressure — Noninvasive respiratory support with continuous positive airway pressure
  Arms: ncpap

SUMMARY:
The purpose of this study is to compare if a new noninvasive ventilation mode (NIV NAVA) is better in noninvasive ventilation of premature infants than currently used Nasal Continuous Airway Pressure (ncpap), and if NIV NAVA gives real benefits for patients or not.

The investigators study hypothesis is that with NIV NAVA the invasive ventilation is more synchronous with patient, which will lead to a decrease in need of inspired oxygen.

ELIGIBILITY:
Inclusion Criteria:

* postconceptional age 28+0 - 36+6
* need of ncpap treatment and inspired oxygen for at least 60 minutes

Exclusion Criteria:

* severe birth asphyxia, malformation or chromosomal abnormality, or other condition, which will decrease life expectancy
* any condition which prevents insertion of naso/orogastric tube

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Duration of inspired oxygen supply | 30minutes- 3weeks
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

SECONDARY OUTCOMES:
Duration of noninvasive ventilation | 30 minutes - 3 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Fraction of inspired oxygen | 0, 1, 3 and 6hours, after which every 6 hours
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Blood gas analyses | 3 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks.
Duration of parenteral nutrition | 3 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University hospital, Oulu, Finland